CLINICAL TRIAL: NCT05336123
Title: The Peace of Mind and Body Project: Treatment Development of Yoga for Anger Management in Incarcerated Adults
Acronym: POMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Butler Hospital (Other); The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1811002261; 5R34AT010172 (NIH)
Record Dates: First submitted 2022-03-31; First posted 2022-04-20 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Anger; Aggression
Keywords: Yoga; Health Education; Aggression; Anger; Incarceration
MeSH Terms: conditions — Aggression; Health Education

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either a 10 week hatha yoga class or health education class.
Who Masked: Investigator
Masking Description: One of the study MPIs and all but one of the Co-Investigators will be blind to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hatha Yoga (Experimental): Participants will be invited to attend one 60-75 minute yoga class for 10 weeks in the prison facility where they reside. Each class will consist of: breathing exercises, brief guided centering meditation, warm-ups, standing postures, floor postures, an inversion, relaxation, and between-class practice assignments. Classes will emphasize mindfulness, including noticing emotions, thoughts, and physical sensations related to anger, and moderate physical activity. Classes will include some teaching of a relevant yoga theme, such as nonviolence (ahimsa).
  Interventions: Behavioral: Hatha Yoga
- Health Education (Active Comparator): To match for attention, the control condition will be a 10-week program that consists of weekly 60-75 minute group classes. In classes, instructors will provide information about general health topics through a variety of means such as slides and handouts. There will be an emphasis on group discussion of relevant topics; instructors do not just lecture. The core rationale for this course is that good physical health is important for good mental health. Instructors will provide information and encourage questions but avoid psychotherapeutic techniques or personalized goal-setting. Instructors will give participants readings to explore on their own.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Hatha Yoga — Weekly hatha yoga classes lasting 10 weeks.
  Arms: Hatha Yoga
Behavioral: Health Education — Weekly health education classes lasting 10 weeks.
  Arms: Health Education

SUMMARY:
The investigators will conduct a pilot randomized clinical trial (n = 40) of hatha yoga vs. a health education group (attention control) for prisoners high in self-reported anger dysregulation. The investigators will assess feasibility and acceptability of the yoga program, the health education control group, and research procedures.

DETAILED DESCRIPTION:
In the criminal justice (CJ) system in the US, there are high rates of mental health and substance use disorders. Although prisons must provide treatment, the CJ system is resource-poor and the presenting problems of prisoners are diverse. To maximize efficiency in the CJ context, recent efforts focus adjunctive interventions on symptoms that are most detrimental to prisoners, and that are shared across diverse conditions. Of particular interest has been anger dysregulation, as this is prevalent in CJ-involved populations, contributing not only to distress and exacerbation of other mental health problems, but also to risk of aggression. Overt aggression further increases risk for prison behavioral infractions or placement in restraints or seclusion, and may delay parole or release decisions.

There are many limitations to existing approaches to anger management in prison. The investigators propose that hatha yoga could serve as a useful adjunctive treatment for anger within prisons. In addition to preliminary research showing that yoga programs may improve anger regulation, research has also demonstrated benefits of yoga for related symptoms of depression, anxiety, and trauma-related emotion reactivity and arousal. Yoga may be delivered in a relatively low-cost fashion. Finally, prisoners may view yoga as less stigmatizing than more traditional anger management interventions, particularly given its focus on physical body awareness/movement and on overall wellness.

Despite a recent proliferation of yoga programs for various problems in prisons, empirical research on this topic is minimal, with a small number of studies limited by significant methodological concerns. The investigators propose to conduct systematic treatment development research that would prepare us to study whether yoga (vs. a health education control group) is an effective adjunctive treatment for prisoners with anger dysregulation.

The investigators will conduct a pilot randomized clinical trial (n = 40) of hatha yoga vs. a health education group (attention control) for prisoners high in self-reported anger dysregulation. Participants will be enrolled in the active intervention for 10 weeks, and then followed for 8 weeks. The investigators will assess feasibility and acceptability of the yoga program, the health education control group, and research procedures. To assess safety, they will track all adverse events in a structured fashion. The investigators will iteratively revise manuals and materials, making final revisions at the end of the pilot RCT. If successful, this project will provide us with materials, experience, and pilot data needed for the next stage of this line of research, namely, a fully powered RCT.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Clinically significant anger dysregulation, as evidenced by a score ≥ 86 on the Novaco Anger Scale (NAS)
* Prisoner or jail detainee, with anticipated duration of remaining time incarcerated of 90 days or more, allowing for participation in the 10 week intervention
* Ability and willingness to provide informed consent
* Willingness to be audio recorded in the intervention condition sessions (e.g., yoga or health education groups).

Exclusion Criteria:

* Presence of current manic or psychotic symptoms, or suicide risk (warranting referral to prison mental health clinical staff)
* Any endorsed item on the Physical Activity Readiness Questionnaire (PAR-Q) except for item 6 (i.e., participants can be included even if they endorse item 6)
* Current weekly yoga practice or current participation in mindfulness- based programming
* Pregnancy
* Inability to understand English sufficiently well to understand the consent form or assessment instruments when read aloud.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-12 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M Weinstock, PhD, Principal Investigator — Brown University
Locations (1):
- Rhode Island Department of Corrections, Cranston, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uebelacker LA, Stevens L, Graves H, Braun TD, Foster R, Johnson JE, Tremont G, Weinstock LM. Pilot Randomized Controlled Trial of a Yoga-Based Intervention Targeting Anger Management for People Who Are Incarcerated. J Integr Complement Med. 2025 Feb;31(2):183-195. doi: 10.1089/jicm.2024.0308. Epub 2024 Oct 7. PMID 39373144

RESULTS

PARTICIPANT FLOW:
Groups:
- Hatha Yoga: 10 weeks of hatha yoga.
  Yoga: Hatha yoga for incarcerated adults.
- Health Education: 10 weeks of Heath Education
  Health Education: Health Education classes for incarcerated adults.
Period: Overall Study
Arm/Group | Hatha Yoga | Health Education
Started | 20 | 20
Completed | 18 | 19
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Hatha Yoga: 10 weeks of hatha yoga
  Yoga: Hatha yoga for incarcerated adults
- Health Education: 10 weeks of health education
  Health Education: Health education classes for incarcerated adults
- Total: Total of all reporting groups
Arm/Group | Hatha Yoga | Health Education | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.85 (6.52) | 33.35 (8.88) | 32.10 (7.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 14 | 15 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 10 | 12 | 22
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Program Satisfaction
Description: Program Satisfaction as measured by the Client Satisfaction Questionnaire (CSQ-8) total score. The CSQ-8 is an 8-item measure with each item measured on a 1-4 scale. Items are summed, with a total score range from 8-32. Higher scores indicate greater client satisfaction.
Time Frame: Assessed at the end of the program (hatha yoga or health education) at week 10
Population: Results for this outcome are reported for the 34 participants of 40 randomized who completed this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga | Health Education
Number analyzed (Participants) | 17 | 17
score on a scale | 29.76 (3.09) | 26.69 (4.01)

2. Secondary Outcome: Program Credibility
Description: Credibility as assessed by Credibility Expectancy Questionnaire (CEQ), credibility subscale. The credibility subscale of the CEQ consists of 3 items from the 6 item CEQ. The 3 items are scored on a range of 0-1, and the mean of these is used in analysis. Higher scores indicate greater intervention credibility.
Time Frame: Assessed at beginning of the program at week 1
Population: Results for this outcome are reported for the 37 participants of 40 randomized who completed this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga | Health Education
Number analyzed (Participants) | 19 | 18
score on a scale | 0.86 (0.13) | 0.81 (0.13)

3. Secondary Outcome: Program Expectancy
Description: Expectancy assessed with the Credibility Expectancy Questionnaire (CEQ), expectancy subscale. The expectancy subscale is a 3 item subscale of the 6 item CEQ. The 3 items are each scored on a range of 0-1, and the mean of of this is used in analysis. Higher scores indicate greater expectations that the intervention will be beneficial.
Time Frame: Assessed at beginning of the program at week 1
Population: Results for this outcome are reported for the 37 participants of 40 randomized who completed this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga | Health Education
Number analyzed (Participants) | 19 | 18
score on a scale | 0.76 (0.18) | 0.67 (0.21)

4. Secondary Outcome: Class Attendance
Description: Number of participants who met class attendance target (6/10 classes total) as assessed through weekly attendance ratings.
Time Frame: Assessed at each weekly class for 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Hatha Yoga | Health Education
Number analyzed (Participants) | 20 | 20
Participants | 10 | 12

5. Secondary Outcome: Novaco Anger Scale
Description: Anger severity was assessed using the Novaco Anger Scale (NAS) from the Novaco Anger Scale and Provocation Inventory (NAS-PI). The NAS is a 48 item measure with each item rated from 1-3. Items are summed, with scores that range from 48-144. Higher scores are indicative of greater experiences of anger. For this study, we report average change in scores from the baseline to the 10 week-follow-up, upon completion of the study intervention. Hence, a positive (vs. negative) change score reflects a reduction in anger from baseline to 10 week follow-up. Higher change scores reflect larger reductions in anger severity.
Time Frame: Change from baseline to the 10 week follow-up
Population: Of the 40 participants randomized, 31 (n=15 in Hatha Yoga; n=16 in Health Education) completed the NAS at the follow-up assessment time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga | Health Education
Number analyzed (Participants) | 15 | 16
score on a scale | 11.87 (14.32) | 5.94 (9.84)

ADVERSE EVENTS:
Time Frame: The period from baseline to the 10 week follow-up
Arm/Group | Hatha Yoga | Health Education
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hatha Yoga (N=20) | Health Education (N=20)
Non-serious adverse event possibly related to study participation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — One participant in the hatha yoga arm reported new back pain; they did not believe it was related to yoga but the investigators judged it to be "possibly" related simply because it occurred during the time period they were taking yoga classes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT05336123/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT05336123/ICF_000.pdf